CLINICAL TRIAL: NCT03608891
Title: Patient Specific Three-Dimensional Titanium Plates Versus Conventional Miniplates for Treatment of Mandibular Body Fractures. (Randomized Clinical Trial)
Brief Title: Patient Specific Plates Versus Conventional Miniplates for Treatment of Mandibular Body Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Adel, Master degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Patient specific plate
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Conventional titanium miniplates
  Interventions: Device: Conventional titanium miniplates
- Intervention arm (Experimental): Patient specific 3D plates
  Interventions: Device: Computer guided patient specific 3D titanium plate

INTERVENTIONS:
Device: Computer guided patient specific 3D titanium plate — CBCT or CT scan will be done preoperatively and dicom files will be imported to mimics software to design and print the patient specific 3D titanium plate.
  Other Names: Intervention Arm
  Arms: Intervention arm
Device: Conventional titanium miniplates — In this group two miniplates of titanium Mini-System 2.0 mm will be used. The plate has profile height 1.0 mm whereas the screw length varies according to the site of the plate. According to Champy osteosynthesis lines for fixation of the posterior mandibular fracture ,the first plate will be placed at the inferior border from the buccal side, using bicortical screws engaging the buccal and lingual cortices to achieve rigid fixation, while the second plate will be placed at about 5mm superior to the inferior plate in the subapical region, using monocortical screws engaging only the buccal cortex to avoid injuring the teeth roots.
  Other Names: Control arm
  Arms: Control Arm

SUMMARY:
The aim of the current study is to evaluate and assess the clinical stability and efficacy of patient specific computer guided titanium plates versus the conventional titanium mini plates regarding accurate reduction and fixation of mandibular body fractures, reducing the operating time, achieving precise bone alignment and reducing the plate palpability.

DETAILED DESCRIPTION:
The study will be conducted on two groups:

Intervention group: patient specific three-dimensional titanium plates CBCT or CT scan will be performed for the patient, the dicom files will be imported into a surgical planning software , plates will then be designed virtually and sent for three-dimensional (3D) printing.

Control group: Conventional miniplates:

In this group two miniplates of titanium Mini-System 2.0 mm will be used. The plate has profile height 1.0 mm whereas the screw length varies according to the site of the plate. According to Champy osteosynthesis lines for fixation of the posterior mandibular fracture ,the first plate will be placed at the inferior border from the buccal side, using bicortical screws engaging the buccal and lingual cortices to achieve rigid fixation, while the second plate will be placed at about 5mm superior to the inferior plate in the subapical region, using monocortical screws engaging only the buccal cortex to avoid injuring the teeth roots.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral mandibular body fractures, not associated with other mandibular and maxillofacial fractures

Exclusion Criteria:

* Patients with bilateral mandibular fractures
* Patients with other mandibular or maxillofacial fractures
* Comminuted fractures
* Medical problem that may interfere with the procedure such as bleeding disorder and pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction measured with visual analogue scale (0-10) | Measured immediately after the surgery
  patient satisfaction is defined as patient-reported outcome measure while the structures and processes of care can be measured by patient-reported experiences (30). Measured on a visual analogue scale (VAS) (29) of 0-10 ,with zero being unsatisfied and 10 being satisfied. Patient Satisfaction is assessed regarding prescence of pain, occlusal discrepencies and overall patient satisfaction.

SECONDARY OUTCOMES:
Fracture gap distance | 0 and 3 months
  This is done using CBCT through measuring the fracture gap distance in millimeters to evaluate proper reduction and fixation
Occlusal bite force | 0 and 3 months
  The biting force will be measured through the follow up visits (1 week,3 months) by the bite force recorder at the incisor region, right and left molar region. The measurement of the bite force will be undertaken using a portable type of occlusal force gauge (GM10, Nagano Keiki, Japan) called OCCLUSAL FORCE-METER GM10. (36)
Operating time | time of the surgery
  The time of the surgery will be recorded using a stopwatch.
Plate palpability | 0 and 3 months
  Measured during all follow up visits, by questioning the patient ,where the patient will be informed of the site of the plates ,and asked if he feels the plates are palpable ,and will be measured by binary measuring unit (yes/no) , also the plates will be palpated by the operator at follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Farid, PHD, Principal Investigator — Cairo University; Mohamed A Abd el Rasol, PhD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez R, Oeltjen JC, Thaller SR. A review of mandibular angle fractures. Craniomaxillofac Trauma Reconstr. 2011 Jun;4(2):69-72. doi: 10.1055/s-0031-1272903. PMID 22655117
- [Background] Goiato MC, Santos MR, Pesqueira AA, Moreno A, dos Santos DM, Haddad MF. Prototyping for surgical and prosthetic treatment. J Craniofac Surg. 2011 May;22(3):914-7. doi: 10.1097/SCS.0b013e31820f7f90. PMID 21558926
- [Background] Levine JP, Patel A, Saadeh PB, Hirsch DL. Computer-aided design and manufacturing in craniomaxillofacial surgery: the new state of the art. J Craniofac Surg. 2012 Jan;23(1):288-93. doi: 10.1097/SCS.0b013e318241ba92. PMID 22337427
- [Background] Talwar RM, Chemaly D. Information and computer technology in oral and maxillofacial surgery. Oral Maxillofac Surg Clin North Am. 2008 Feb;20(1):79-89. doi: 10.1016/j.coms.2007.09.006. PMID 18194740
- [Background] Edwards SP. Computer-assisted craniomaxillofacial surgery. Oral Maxillofac Surg Clin North Am. 2010 Feb;22(1):117-34. doi: 10.1016/j.coms.2009.11.005. PMID 20159482
- [Background] Hassfeld S, Muhling J. Computer assisted oral and maxillofacial surgery--a review and an assessment of technology. Int J Oral Maxillofac Surg. 2001 Feb;30(1):2-13. doi: 10.1054/ijom.2000.0024. PMID 11289616
- [Background] Eckardt A, Swennen GR. Virtual planning of composite mandibular reconstruction with free fibula bone graft. J Craniofac Surg. 2005 Nov;16(6):1137-40. doi: 10.1097/01.scs.0000186306.32042.96. PMID 16327572
- [Background] Bell RB. Computer planning and intraoperative navigation in cranio-maxillofacial surgery. Oral Maxillofac Surg Clin North Am. 2010 Feb;22(1):135-56. doi: 10.1016/j.coms.2009.10.010. PMID 20159483
- [Result] Al-Abri R, Al-Balushi A. Patient satisfaction survey as a tool towards quality improvement. Oman Med J. 2014 Jan;29(1):3-7. doi: 10.5001/omj.2014.02. PMID 24501659
- [Result] Butts SC, Floyd E, Lai E, Rosenfeld RM, Doerr T. Reporting of Postoperative Pain Management Protocols in Randomized Clinical Trials of Mandibular Fracture Repair: A Systematic Review. JAMA Facial Plast Surg. 2015 Nov-Dec;17(6):440-8. doi: 10.1001/jamafacial.2015.1011. PMID 26335408
- [Result] Kumar ST, Saraf S, Devi SP. Evaluation of bite force after open reduction and internal fixation using microplates. J Dent (Tehran). 2013 Sep;10(5):466-77. Epub 2013 Sep 30. PMID 24910656
- [Result] Rodt T, Bartling SO, Zajaczek JE, Vafa MA, Kapapa T, Majdani O, Krauss JK, Zumkeller M, Matthies H, Becker H, Kaminsky J. Evaluation of surface and volume rendering in 3D-CT of facial fractures. Dentomaxillofac Radiol. 2006 Jul;35(4):227-31. doi: 10.1259/dmfr/22989395. PMID 16798916
- [Result] Manson PN, Markowitz B, Mirvis S, Dunham M, Yaremchuk M. Toward CT-based facial fracture treatment. Plast Reconstr Surg. 1990 Feb;85(2):202-12; discussion 213-4. PMID 2300626